CLINICAL TRIAL: NCT00011713
Title: Human Exposure to Bisphenol A, Phthalates and Fertility, Pregnancy Outcomes.
Brief Title: Environment and Reproductive Health; Human Exposure to Bisphenol A, Phthalates and Fertility and Pregnancy Outcomes
Acronym: EARTH
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Russ Hauser, Frederick Lee Hisaw Professor of Reproductive Physiology, National Institute of Environmental Health Sciences (NIEHS)
Other Study IDs: ES 009718; 2R01ES009718-16 (NIH)
Record Dates: First submitted 2001-02-27; First posted 2001-03-01 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Infertility
Keywords: Semen; Infertility; ART - Assisted Reproduction Technology; Phthalates; Bisphenol A
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine, semen, follicular fluid, amniotic fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infertility patients: Patients undergoing infertility treatment at Massachusetts General Hospital Infertility Clinic.
  Interventions: Other: Completion questionnaires/providing biological samples

INTERVENTIONS:
Other: Completion questionnaires/providing biological samples — Participant completes baseline interview at enrollment, then completes online questionnaire on lifestyle and medical history. Diet questionnaire is completed at home and mailed back. Online questionnaire about personal care product use and medications is completed at each scheduled study visit.

SUMMARY:
The purpose of the study is to investigate the relationship between environmental agents and reproductive health. Environmental agents of interest include exposure to chemicals such as polychlorinated biphenyls (PCBs), flame retardants, dioxins, bisphenol A, phthalates, pesticides, and metals like lead and cadmium. We are also interested in the relationship between reproductive health and lifestyle risk factors, such as exposure to environmental tobacco smoke. Enrollees are asked to participate in this study because they and their partner are patients of the MGH Fertility Center, trying to get pregnant, either naturally or by undergoing Intrauterine Insemination (IUI) and/or In Vitro Fertilization (IVF).

DETAILED DESCRIPTION:
Specific Aim #1: To determine the association of a mixture of paternal urinary concentrations of phthalate metabolites, BPA and parabens with the primary outcomes of implantation failure and live birth, and the secondary outcomes of chemical pregnancy (with no subsequent clinical pregnancy) and spontaneous abortion.

Hypothesis 1: Higher paternal urinary concentrations of a mixture of anti-androgenic phthalate metabolites of DEHP, DBP, DiBP, BBzP, and DiNP is associated with increased risk of implantation failure and reduced live birth rate, and increased risk of chemical pregnancy and spontaneous abortion.

Hypothesis 2: Higher paternal urinary concentrations of a mixture of estrogenic chemicals (BPA and parabens) is associated with increased risk of implantation failure and reduced live birth rate, and increased risk of chemical pregnancy and spontaneous abortion.

Specific Aim #2: To determine the association of a mixture of maternal urinary concentrations of phthalate metabolites, BPA and parabens with implantation failure and live birth rate, and the secondary outcomes of chemical pregnancy and spontaneous abortion.

Hypothesis 2: Higher maternal urinary concentrations of a mixture of anti-androgenic phthalate metabolites of DEHP, DBP, DiBP, BBzP, and DiNP is associated with increased risk of implantation failure and reduced live birth rate, and increased risk of chemical pregnancy and spontaneous abortion.

Hypothesis 3: Higher maternal urinary concentrations of a mixture of estrogenic BPA and parabens is associated with increased risk of implantation failure and reduced live birth rate, and increased risk of chemical pregnancy and spontaneous abortion.

Specific Aim #3: To determine the joint effect of maternal and paternal urinary concentrations of phthalate metabolites, BPA and parabens with primary outcomes of interest including implantation failure and live birth rate, and the secondary outcomes of chemical pregnancy and spontaneous abortion.

ELIGIBILITY:
Inclusion Criteria:

1. Couples undergoing treatment for infertility at MGH Clinic
2. Men 18-55 years old
3. Women 18 - 45 years old

Exclusion Criteria:

1. Any individual or couple who is not undergoing infertility treatment at MGH Clinic and or who is outside of age range.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study subjects will be recruited from couples seeking treatment of infertility at the MGH IVF Clinic. Men and women must be at least 18 years old to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1474 (Actual)
Dates: Start 1999-10 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Paternal Exposure to Environmental Chemicals | 2019
  To determine the association of a mixture of paternal urinary concentrations of phthalate metabolites, BPA and parabens with the primary outcomes of implantation failure and live birth, and the secondary outcomes of chemical pregnancy (with no subsequent clinical pregnancy) and spontaneous abortion.

SECONDARY OUTCOMES:
Maternal Exposure to Environmental Chemicals | 2019
  To determine the association of a mixture of maternal urinary concentrations of phthalate metabolites, BPA and parabens with implantation failure and live birth rate, and the secondary outcomes of chemical pregnancy and spontaneous abortion.

CONTACTS AND LOCATIONS:
Overall Officials: Russ Hauser, MD, ScD, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States

REFERENCES:
- [Result] Meeker JD, Singh NP, Hauser R. Serum concentrations of estradiol and free T4 are inversely correlated with sperm DNA damage in men from an infertility clinic. J Androl. 2008 Jul-Aug;29(4):379-88. doi: 10.2164/jandrol.107.004416. Epub 2008 Mar 20. PMID 18359755
- [Result] Chavarro JE, Toth TL, Sadio SM, Hauser R. Soy food and isoflavone intake in relation to semen quality parameters among men from an infertility clinic. Hum Reprod. 2008 Nov;23(11):2584-90. doi: 10.1093/humrep/den243. Epub 2008 Jul 23. PMID 18650557
- [Result] Chavarro JE, Toth TL, Wright DL, Meeker JD, Hauser R. Body mass index in relation to semen quality, sperm DNA integrity, and serum reproductive hormone levels among men attending an infertility clinic. Fertil Steril. 2010 May 1;93(7):2222-31. doi: 10.1016/j.fertnstert.2009.01.100. Epub 2009 Mar 3. PMID 19261274
- [Result] Meeker JD, Missmer SA, Altshul L, Vitonis AF, Ryan L, Cramer DW, Hauser R. Serum and follicular fluid organochlorine concentrations among women undergoing assisted reproduction technologies. Environ Health. 2009 Jul 14;8:32. doi: 10.1186/1476-069X-8-32. PMID 19594949
- [Result] Mok-Lin E, Ehrlich S, Williams PL, Petrozza J, Wright DL, Calafat AM, Ye X, Hauser R. Urinary bisphenol A concentrations and ovarian response among women undergoing IVF. Int J Androl. 2010 Apr;33(2):385-93. doi: 10.1111/j.1365-2605.2009.01014.x. Epub 2009 Nov 30. PMID 20002217
- [Result] Meeker JD, Calafat AM, Hauser R. Urinary bisphenol A concentrations in relation to serum thyroid and reproductive hormone levels in men from an infertility clinic. Environ Sci Technol. 2010 Feb 15;44(4):1458-63. doi: 10.1021/es9028292. PMID 20030380
- [Result] Meeker JD, Ehrlich S, Toth TL, Wright DL, Calafat AM, Trisini AT, Ye X, Hauser R. Semen quality and sperm DNA damage in relation to urinary bisphenol A among men from an infertility clinic. Reprod Toxicol. 2010 Dec;30(4):532-9. doi: 10.1016/j.reprotox.2010.07.005. Epub 2010 Jul 23. PMID 20656017
- [Result] Chavarro JE, Furtado J, Toth TL, Ford J, Keller M, Campos H, Hauser R. Trans-fatty acid levels in sperm are associated with sperm concentration among men from an infertility clinic. Fertil Steril. 2011 Apr;95(5):1794-7. doi: 10.1016/j.fertnstert.2010.10.039. Epub 2010 Nov 11. PMID 21071027
- [Result] Braun JM, Smith KW, Williams PL, Calafat AM, Berry K, Ehrlich S, Hauser R. Variability of urinary phthalate metabolite and bisphenol A concentrations before and during pregnancy. Environ Health Perspect. 2012 May;120(5):739-45. doi: 10.1289/ehp.1104139. Epub 2012 Jan 19. PMID 22262702
- [Result] Attaman JA, Toth TL, Furtado J, Campos H, Hauser R, Chavarro JE. Dietary fat and semen quality among men attending a fertility clinic. Hum Reprod. 2012 May;27(5):1466-74. doi: 10.1093/humrep/des065. Epub 2012 Mar 13. PMID 22416013
- [Result] Ehrlich S, Williams PL, Missmer SA, Flaws JA, Berry KF, Calafat AM, Ye X, Petrozza JC, Wright D, Hauser R. Urinary bisphenol A concentrations and implantation failure among women undergoing in vitro fertilization. Environ Health Perspect. 2012 Jul;120(7):978-83. doi: 10.1289/ehp.1104307. Epub 2012 Apr 6. PMID 22484414
- [Result] Chavarro JE, Ehrlich S, Colaci DS, Wright DL, Toth TL, Petrozza JC, Hauser R. Body mass index and short-term weight change in relation to treatment outcomes in women undergoing assisted reproduction. Fertil Steril. 2012 Jul;98(1):109-16. doi: 10.1016/j.fertnstert.2012.04.012. Epub 2012 May 16. PMID 22607889
- [Result] Ferguson KK, Hauser R, Altshul L, Meeker JD. Serum concentrations of p, p'-DDE, HCB, PCBs and reproductive hormones among men of reproductive age. Reprod Toxicol. 2012 Nov;34(3):429-35. doi: 10.1016/j.reprotox.2012.04.006. Epub 2012 May 5. PMID 22564984
- [Result] Meeker JD, Calafat AM, Hauser R. Urinary phthalate metabolites and their biotransformation products: predictors and temporal variability among men and women. J Expo Sci Environ Epidemiol. 2012 Jul;22(4):376-85. doi: 10.1038/jes.2012.7. Epub 2012 Feb 22. PMID 22354176
- [Result] Smith KW, Braun JM, Williams PL, Ehrlich S, Correia KF, Calafat AM, Ye X, Ford J, Keller M, Meeker JD, Hauser R. Predictors and variability of urinary paraben concentrations in men and women, including before and during pregnancy. Environ Health Perspect. 2012 Nov;120(11):1538-43. doi: 10.1289/ehp.1104614. Epub 2012 Jun 21. PMID 22721761
- [Result] Colaci DS, Afeiche M, Gaskins AJ, Wright DL, Toth TL, Tanrikut C, Hauser R, Chavarro JE. Men's body mass index in relation to embryo quality and clinical outcomes in couples undergoing in vitro fertilization. Fertil Steril. 2012 Nov;98(5):1193-9.e1. doi: 10.1016/j.fertnstert.2012.07.1102. Epub 2012 Aug 9. PMID 22884013
- [Result] Ehrlich S, Williams PL, Missmer SA, Flaws JA, Ye X, Calafat AM, Petrozza JC, Wright D, Hauser R. Urinary bisphenol A concentrations and early reproductive health outcomes among women undergoing IVF. Hum Reprod. 2012 Dec;27(12):3583-92. doi: 10.1093/humrep/des328. Epub 2012 Sep 26. PMID 23014629
- [Result] Hernandez-Diaz S, Su YC, Mitchell AA, Kelley KE, Calafat AM, Hauser R. Medications as a potential source of exposure to phthalates among women of childbearing age. Reprod Toxicol. 2013 Jun;37:1-5. doi: 10.1016/j.reprotox.2013.01.001. Epub 2013 Jan 18. PMID 23333816
- [Result] Smith KW, Souter I, Dimitriadis I, Ehrlich S, Williams PL, Calafat AM, Hauser R. Urinary paraben concentrations and ovarian aging among women from a fertility center. Environ Health Perspect. 2013 Nov-Dec;121(11-12):1299-305. doi: 10.1289/ehp.1205350. Epub 2013 Aug 2. PMID 23912598
- [Result] Cantonwine DE, Hauser R, Meeker JD. Bisphenol A and Human Reproductive Health. Expert Rev Obstet Gynecol. 2013 Jul 1;8(4):10.1586/17474108.2013.811939. doi: 10.1586/17474108.2013.811939. PMID 24187577
- [Result] Ehrlich S, Williams PL, Hauser R, Missmer SA, Peretz J, Calafat AM, Flaws JA. Urinary bisphenol A concentrations and cytochrome P450 19 A1 (Cyp19) gene expression in ovarian granulosa cells: an in vivo human study. Reprod Toxicol. 2013 Dec;42:18-23. doi: 10.1016/j.reprotox.2013.06.071. Epub 2013 Jul 10. PMID 23850856
- [Result] Braun JM, Just AC, Williams PL, Smith KW, Calafat AM, Hauser R. Personal care product use and urinary phthalate metabolite and paraben concentrations during pregnancy among women from a fertility clinic. J Expo Sci Environ Epidemiol. 2014 Sep-Oct;24(5):459-66. doi: 10.1038/jes.2013.69. Epub 2013 Oct 23. PMID 24149971
- [Result] Machtinger R, Combelles CM, Missmer SA, Correia KF, Williams P, Hauser R, Racowsky C. Bisphenol-A and human oocyte maturation in vitro. Hum Reprod. 2013 Oct;28(10):2735-45. doi: 10.1093/humrep/det312. Epub 2013 Jul 30. PMID 23904465
- [Result] Souter I, Smith KW, Dimitriadis I, Ehrlich S, Williams PL, Calafat AM, Hauser R. The association of bisphenol-A urinary concentrations with antral follicle counts and other measures of ovarian reserve in women undergoing infertility treatments. Reprod Toxicol. 2013 Dec;42:224-31. doi: 10.1016/j.reprotox.2013.09.008. Epub 2013 Oct 4. PMID 24100206
- [Result] Afeiche MC, Bridges ND, Williams PL, Gaskins AJ, Tanrikut C, Petrozza JC, Hauser R, Chavarro JE. Dairy intake and semen quality among men attending a fertility clinic. Fertil Steril. 2014 May;101(5):1280-7. doi: 10.1016/j.fertnstert.2014.02.003. Epub 2014 Mar 14. PMID 24636397
- [Result] Afeiche MC, Gaskins AJ, Williams PL, Toth TL, Wright DL, Tanrikut C, Hauser R, Chavarro JE. Processed meat intake is unfavorably and fish intake favorably associated with semen quality indicators among men attending a fertility clinic. J Nutr. 2014 Jul;144(7):1091-8. doi: 10.3945/jn.113.190173. Epub 2014 May 21. PMID 24850626
- [Result] Gaskins AJ, Afeiche MC, Hauser R, Williams PL, Gillman MW, Tanrikut C, Petrozza JC, Chavarro JE. Paternal physical and sedentary activities in relation to semen quality and reproductive outcomes among couples from a fertility center. Hum Reprod. 2014 Nov;29(11):2575-82. doi: 10.1093/humrep/deu212. Epub 2014 Aug 27. PMID 25164027
- [Result] Gaskins AJ, Afeiche MC, Wright DL, Toth TL, Williams PL, Gillman MW, Hauser R, Chavarro JE. Dietary folate and reproductive success among women undergoing assisted reproduction. Obstet Gynecol. 2014 Oct;124(4):801-809. doi: 10.1097/AOG.0000000000000477. PMID 25198264
- [Result] Minguez-Alarcon L, Afeiche MC, Williams PL, Arvizu M, Tanrikut C, Amarasiriwardena CJ, Ford JB, Hauser R, Chavarro JE; Earth Study Team. Hair mercury (Hg) levels, fish consumption and semen parameters among men attending a fertility center. Int J Hyg Environ Health. 2018 Mar;221(2):174-182. doi: 10.1016/j.ijheh.2017.10.014. Epub 2017 Oct 28. PMID 29102416
- [Result] Messerlian C, Mustieles V, Minguez-Alarcon L, Ford JB, Calafat AM, Souter I, Williams PL, Hauser R; Environment and Reproductive Health (EARTH) Study Team. Preconception and prenatal urinary concentrations of phenols and birth size of singleton infants born to mothers and fathers from the Environment and Reproductive Health (EARTH) study. Environ Int. 2018 May;114:60-68. doi: 10.1016/j.envint.2018.02.017. Epub 2018 Feb 22. PMID 29477955
- [Result] Chiu YH, Williams PL, Gillman MW, Gaskins AJ, Minguez-Alarcon L, Souter I, Toth TL, Ford JB, Hauser R, Chavarro JE; EARTH Study Team. Association Between Pesticide Residue Intake From Consumption of Fruits and Vegetables and Pregnancy Outcomes Among Women Undergoing Infertility Treatment With Assisted Reproductive Technology. JAMA Intern Med. 2018 Jan 1;178(1):17-26. doi: 10.1001/jamainternmed.2017.5038. PMID 29084307
- [Result] Chiu YH, Karmon AE, Gaskins AJ, Arvizu M, Williams PL, Souter I, Rueda BR, Hauser R, Chavarro JE; EARTH Study Team. Serum omega-3 fatty acids and treatment outcomes among women undergoing assisted reproduction. Hum Reprod. 2018 Jan 1;33(1):156-165. doi: 10.1093/humrep/dex335. PMID 29136189
- [Result] Segal TR, Minguez-Alarcon L, Chiu YH, Williams PL, Nassan FL, Dadd R, Ospina M, Calafat AM, Hauser R; Earth Study Team. Urinary concentrations of 3-(diethylcarbamoyl)benzoic acid (DCBA), a major metabolite of N,N-diethyl-m-toluamide (DEET) and semen parameters among men attending a fertility center. Hum Reprod. 2017 Dec 1;32(12):2532-2539. doi: 10.1093/humrep/dex327. PMID 29077936
- [Result] Messerlian C, Mustieles V, Wylie BJ, Ford JB, Keller M, Ye X, Calafat AM, Williams PL, Hauser R; Environment Team Reproductive Health Study. Ultrasound gel as an unrecognized source of exposure to phthalates and phenols among pregnant women undergoing routine scan. Int J Hyg Environ Health. 2017 Nov;220(8):1285-1294. doi: 10.1016/j.ijheh.2017.08.003. Epub 2017 Aug 14. PMID 28830670
- [Result] Messerlian C, Braun JM, Minguez-Alarcon L, Williams PL, Ford JB, Mustieles V, Calafat AM, Souter I, Toth T, Hauser R; Environment and Reproductive Health (EARTH) Study Team. Paternal and maternal urinary phthalate metabolite concentrations and birth weight of singletons conceived by subfertile couples. Environ Int. 2017 Oct;107:55-64. doi: 10.1016/j.envint.2017.06.015. Epub 2017 Jun 27. PMID 28666241
- [Result] Messerlian C, Bellinger D, Minguez-Alarcon L, Romano ME, Ford JB, Williams PL, Calafat AM, Hauser R, Braun JM. Paternal and maternal preconception urinary phthalate metabolite concentrations and child behavior. Environ Res. 2017 Oct;158:720-728. doi: 10.1016/j.envres.2017.07.032. Epub 2017 Jul 21. PMID 28738300
- [Result] Souter I, Chiu YH, Batsis M, Afeiche MC, Williams PL, Hauser R, Chavarro JE; EARTH Study Team. The association of protein intake (amount and type) with ovarian antral follicle counts among infertile women: results from the EARTH prospective study cohort. BJOG. 2017 Sep;124(10):1547-1555. doi: 10.1111/1471-0528.14630. Epub 2017 Apr 10. PMID 28278351
- [Result] Abadia L, Chiu YH, Williams PL, Toth TL, Souter I, Hauser R, Chavarro JE, Gaskins AJ; EARTH Study Team. The association between pre-treatment maternal alcohol and caffeine intake and outcomes of assisted reproduction in a prospectively followed cohort. Hum Reprod. 2017 Sep 1;32(9):1846-1854. doi: 10.1093/humrep/dex237. PMID 28854726
- [Result] Carignan CC, Minguez-Alarcon L, Butt CM, Williams PL, Meeker JD, Stapleton HM, Toth TL, Ford JB, Hauser R; EARTH Study Team. Urinary Concentrations of Organophosphate Flame Retardant Metabolites and Pregnancy Outcomes among Women Undergoing in Vitro Fertilization. Environ Health Perspect. 2017 Aug 25;125(8):087018. doi: 10.1289/EHP1021. PMID 28858831
- [Result] Minguez-Alarcon L, Christou G, Messerlian C, Williams PL, Carignan CC, Souter I, Ford JB, Calafat AM, Hauser R; EARTH Study Team. Urinary triclosan concentrations and diminished ovarian reserve among women undergoing treatment in a fertility clinic. Fertil Steril. 2017 Aug;108(2):312-319. doi: 10.1016/j.fertnstert.2017.05.020. Epub 2017 Jun 2. PMID 28583664
- [Result] Tiseo BC, Gaskins AJ, Hauser R, Chavarro JE, Tanrikut C; EARTH Study Team. Coenzyme Q10 Intake From Food and Semen Parameters in a Subfertile Population. Urology. 2017 Apr;102:100-105. doi: 10.1016/j.urology.2016.11.022. Epub 2016 Nov 22. PMID 27888150
- [Result] Chiu YH, Minguez-Alarcon L, Ford JB, Keller M, Seely EW, Messerlian C, Petrozza J, Williams PL, Ye X, Calafat AM, Hauser R, James-Todd T; for EARTH Study Team. Trimester-Specific Urinary Bisphenol A Concentrations and Blood Glucose Levels Among Pregnant Women From a Fertility Clinic. J Clin Endocrinol Metab. 2017 Apr 1;102(4):1350-1357. doi: 10.1210/jc.2017-00022. PMID 28323984
- [Result] Karmon AE, Toth TL, Chiu YH, Gaskins AJ, Tanrikut C, Wright DL, Hauser R, Chavarro JE; Earth Study Team. Male caffeine and alcohol intake in relation to semen parameters and in vitro fertilization outcomes among fertility patients. Andrology. 2017 Mar;5(2):354-361. doi: 10.1111/andr.12310. Epub 2017 Feb 10. PMID 28187518
- [Result] Lewis RC, Minguez-Alarcon L, Meeker JD, Williams PL, Mezei G, Ford JB, Hauser R; EARTH Study Team. Self-reported mobile phone use and semen parameters among men from a fertility clinic. Reprod Toxicol. 2017 Jan;67:42-47. doi: 10.1016/j.reprotox.2016.11.008. Epub 2016 Nov 9. PMID 27838386
- [Result] Vanegas JC, Chavarro JE, Williams PL, Ford JB, Toth TL, Hauser R, Gaskins AJ. Discrete survival model analysis of a couple's smoking pattern and outcomes of assisted reproduction. Fertil Res Pract. 2017;3:5. doi: 10.1186/s40738-017-0032-2. Epub 2017 Feb 20. PMID 28480049
- [Result] Lewis RC, Hauser R, Maynard AD, Neitzel RL, Wang L, Kavet R, Morey P, Ford JB, Meeker JD; Earth Study Team. PERSONAL MEASURES OF POWER-FREQUENCY MAGNETIC FIELD EXPOSURE AMONG MEN FROM AN INFERTILITY CLINIC: DISTRIBUTION, TEMPORAL VARIABILITY AND CORRELATION WITH THEIR FEMALE PARTNERS' EXPOSURE. Radiat Prot Dosimetry. 2016 Dec;172(4):401-408. doi: 10.1093/rpd/ncv515. Epub 2015 Dec 24. PMID 26705359
- [Result] Minguez-Alarcon L, Souter I, Chiu YH, Williams PL, Ford JB, Ye X, Calafat AM, Hauser R; Earth Study Team. Urinary concentrations of cyclohexane-1,2-dicarboxylic acid monohydroxy isononyl ester, a metabolite of the non-phthalate plasticizer di(isononyl)cyclohexane-1,2-dicarboxylate (DINCH), and markers of ovarian response among women attending a fertility center. Environ Res. 2016 Nov;151:595-600. doi: 10.1016/j.envres.2016.08.012. Epub 2016 Sep 2. PMID 27591839
- [Result] Messerlian C, Wylie BJ, Minguez-Alarcon L, Williams PL, Ford JB, Souter IC, Calafat AM, Hauser R; Earth Study Team. Urinary Concentrations of Phthalate Metabolites and Pregnancy Loss Among Women Conceiving with Medically Assisted Reproduction. Epidemiology. 2016 Nov;27(6):879-88. doi: 10.1097/EDE.0000000000000525. PMID 27299194
- [Result] Gaskins AJ, Williams PL, Keller MG, Souter I, Hauser R, Chavarro JE; EARTH Study Team. Maternal physical and sedentary activities in relation to reproductive outcomes following IVF. Reprod Biomed Online. 2016 Oct;33(4):513-521. doi: 10.1016/j.rbmo.2016.07.002. Epub 2016 Jul 20. PMID 27474489
- [Result] Minguez-Alarcon L, Gaskins AJ, Chiu YH, Souter I, Williams PL, Calafat AM, Hauser R, Chavarro JE; EARTH Study team. Dietary folate intake and modification of the association of urinary bisphenol A concentrations with in vitro fertilization outcomes among women from a fertility clinic. Reprod Toxicol. 2016 Oct;65:104-112. doi: 10.1016/j.reprotox.2016.07.012. Epub 2016 Jul 14. PMID 27423903
- [Result] Minguez-Alarcon L, Hauser R, Gaskins AJ. Effects of bisphenol A on male and couple reproductive health: a review. Fertil Steril. 2016 Sep 15;106(4):864-70. doi: 10.1016/j.fertnstert.2016.07.1118. Epub 2016 Aug 4. PMID 27498136
- [Result] Abadia L, Gaskins AJ, Chiu YH, Williams PL, Keller M, Wright DL, Souter I, Hauser R, Chavarro JE; Environment and Reproductive Health Study Team. Serum 25-hydroxyvitamin D concentrations and treatment outcomes of women undergoing assisted reproduction. Am J Clin Nutr. 2016 Sep;104(3):729-35. doi: 10.3945/ajcn.115.126359. Epub 2016 Jul 27. PMID 27465382
- [Result] Hu Y, Chiu YH, Hauser R, Chavarro J, Sun Q. Overall and class-specific scores of pesticide residues from fruits and vegetables as a tool to rank intake of pesticide residues in United States: A validation study. Environ Int. 2016 Jul-Aug;92-93:294-300. doi: 10.1016/j.envint.2016.04.028. Epub 2016 Apr 26. PMID 27128714
- [Result] Gaskins AJ, Chiu YH, Williams PL, Keller MG, Toth TL, Hauser R, Chavarro JE; EARTH Study Team. Maternal whole grain intake and outcomes of in vitro fertilization. Fertil Steril. 2016 Jun;105(6):1503-1510.e4. doi: 10.1016/j.fertnstert.2016.02.015. Epub 2016 Feb 28. PMID 26926253
- [Result] Hauser R, Gaskins AJ, Souter I, Smith KW, Dodge LE, Ehrlich S, Meeker JD, Calafat AM, Williams PL; EARTH Study Team. Urinary Phthalate Metabolite Concentrations and Reproductive Outcomes among Women Undergoing in Vitro Fertilization: Results from the EARTH Study. Environ Health Perspect. 2016 Jun;124(6):831-9. doi: 10.1289/ehp.1509760. Epub 2015 Nov 6. PMID 26545148
- [Result] Xia W, Chiu YH, Afeiche MC, Williams PL, Ford JB, Tanrikut C, Souter I, Hauser R, Chavarro JE; EARTH study team. Impact of men's dairy intake on assisted reproductive technology outcomes among couples attending a fertility clinic. Andrology. 2016 Mar;4(2):277-83. doi: 10.1111/andr.12151. Epub 2016 Jan 29. PMID 26825777
- [Result] Chavarro JE, Minguez-Alarcon L, Chiu YH, Gaskins AJ, Souter I, Williams PL, Calafat AM, Hauser R; EARTH Study Team. Soy Intake Modifies the Relation Between Urinary Bisphenol A Concentrations and Pregnancy Outcomes Among Women Undergoing Assisted Reproduction. J Clin Endocrinol Metab. 2016 Mar;101(3):1082-90. doi: 10.1210/jc.2015-3473. Epub 2016 Jan 27. PMID 26815879
- [Result] Afeiche MC, Chiu YH, Gaskins AJ, Williams PL, Souter I, Wright DL, Hauser R, Chavarro JE; EARTH Study team. Dairy intake in relation to in vitro fertilization outcomes among women from a fertility clinic. Hum Reprod. 2016 Mar;31(3):563-71. doi: 10.1093/humrep/dev344. Epub 2016 Jan 18. PMID 26787645
- [Result] Minguez-Alarcon L, Chiu YH, Messerlian C, Williams PL, Sabatini ME, Toth TL, Ford JB, Calafat AM, Hauser R; EARTH Study Team. Urinary paraben concentrations and in vitro fertilization outcomes among women from a fertility clinic. Fertil Steril. 2016 Mar;105(3):714-721. doi: 10.1016/j.fertnstert.2015.11.021. Epub 2015 Dec 2. PMID 26654974
- [Result] Lewis RC, Hauser R, Wang L, Kavet R, Meeker JD. Personal power-frequency magnetic field exposure in women recruited at an infertility clinic: association with physical activity and temporal variability. Radiat Prot Dosimetry. 2016 Mar;168(4):478-88. doi: 10.1093/rpd/ncv365. Epub 2015 Jul 7. PMID 26152565
- [Result] Messerlian C, Souter I, Gaskins AJ, Williams PL, Ford JB, Chiu YH, Calafat AM, Hauser R; Earth Study Team. Urinary phthalate metabolites and ovarian reserve among women seeking infertility care. Hum Reprod. 2016 Jan;31(1):75-83. doi: 10.1093/humrep/dev292. Epub 2015 Nov 15. PMID 26573529
- [Result] Braun JM, Gennings C, Hauser R, Webster TF. What Can Epidemiological Studies Tell Us about the Impact of Chemical Mixtures on Human Health? Environ Health Perspect. 2016 Jan;124(1):A6-9. doi: 10.1289/ehp.1510569. PMID 26720830
- [Result] Lewis RC, Hauser R, Maynard AD, Neitzel RL, Wang L, Kavet R, Meeker JD. Exposure to Power-Frequency Magnetic Fields and the Risk of Infertility and Adverse Pregnancy Outcomes: Update on the Human Evidence and Recommendations for Future Study Designs. J Toxicol Environ Health B Crit Rev. 2016;19(1):29-45. doi: 10.1080/10937404.2015.1134370. PMID 27030583
- [Result] Dodge LE, Williams PL, Williams MA, Missmer SA, Souter I, Calafat AM, Hauser R; EARTH Study Team. Associations between paternal urinary phthalate metabolite concentrations and reproductive outcomes among couples seeking fertility treatment. Reprod Toxicol. 2015 Dec;58:184-93. doi: 10.1016/j.reprotox.2015.09.007. Epub 2015 Oct 9. PMID 26456810
- [Result] Styer AK, Gaskins AJ, Brady PC, Sluss PM, Chavarro JE, Hauser RB, Toth TL. Dynamic antimullerian hormone levels during controlled ovarian hyperstimulation predict in vitro fertilization response and pregnancy outcomes. Fertil Steril. 2015 Nov;104(5):1153-61.e1-7. doi: 10.1016/j.fertnstert.2015.07.1161. Epub 2015 Aug 24. PMID 26315051
- [Result] Gaskins AJ, Chiu YH, Williams PL, Ford JB, Toth TL, Hauser R, Chavarro JE; EARTH Study Team. Association between serum folate and vitamin B-12 and outcomes of assisted reproductive technologies. Am J Clin Nutr. 2015 Oct;102(4):943-50. doi: 10.3945/ajcn.115.112185. Epub 2015 Sep 9. PMID 26354529
- [Result] Xia W, Chiu YH, Williams PL, Gaskins AJ, Toth TL, Tanrikut C, Hauser R, Chavarro JE. Men's meat intake and treatment outcomes among couples undergoing assisted reproduction. Fertil Steril. 2015 Oct;104(4):972-979. doi: 10.1016/j.fertnstert.2015.06.037. Epub 2015 Jul 20. PMID 26206344
- [Result] Minguez-Alarcon L, Gaskins AJ, Chiu YH, Williams PL, Ehrlich S, Chavarro JE, Petrozza JC, Ford JB, Calafat AM, Hauser R; EARTH Study Team. Urinary bisphenol A concentrations and association with in vitro fertilization outcomes among women from a fertility clinic. Hum Reprod. 2015 Sep;30(9):2120-8. doi: 10.1093/humrep/dev183. Epub 2015 Jul 24. PMID 26209788
- [Result] Minguez-Alarcon L, Afeiche MC, Chiu YH, Vanegas JC, Williams PL, Tanrikut C, Toth TL, Hauser R, Chavarro JE. Male soy food intake was not associated with in vitro fertilization outcomes among couples attending a fertility center. Andrology. 2015 Jul;3(4):702-8. doi: 10.1111/andr.12046. Epub 2015 Jun 20. PMID 26097060
- [Result] Dodge LE, Williams PL, Williams MA, Missmer SA, Toth TL, Calafat AM, Hauser R. Paternal Urinary Concentrations of Parabens and Other Phenols in Relation to Reproductive Outcomes among Couples from a Fertility Clinic. Environ Health Perspect. 2015 Jul;123(7):665-71. doi: 10.1289/ehp.1408605. Epub 2015 Mar 13. PMID 25767892
- [Result] Chiu YH, Afeiche MC, Gaskins AJ, Williams PL, Petrozza JC, Tanrikut C, Hauser R, Chavarro JE. Fruit and vegetable intake and their pesticide residues in relation to semen quality among men from a fertility clinic. Hum Reprod. 2015 Jun;30(6):1342-51. doi: 10.1093/humrep/dev064. Epub 2015 Mar 30. PMID 25824023
- [Result] Dodge LE, Kelley KE, Williams PL, Williams MA, Hernandez-Diaz S, Missmer SA, Hauser R. Medications as a source of paraben exposure. Reprod Toxicol. 2015 Apr;52:93-100. doi: 10.1016/j.reprotox.2015.02.002. Epub 2015 Feb 26. PMID 25728410
- [Result] Vanegas JC, Afeiche MC, Gaskins AJ, Minguez-Alarcon L, Williams PL, Wright DL, Toth TL, Hauser R, Chavarro JE. Soy food intake and treatment outcomes of women undergoing assisted reproductive technology. Fertil Steril. 2015 Mar;103(3):749-55.e2. doi: 10.1016/j.fertnstert.2014.12.104. Epub 2015 Jan 7. PMID 25577465
- [Result] Wright DL, Afeiche MC, Ehrlich S, Smith K, Williams PL, Chavarro JE, Batsis M, Toth TL, Hauser R. Hair mercury concentrations and in vitro fertilization (IVF) outcomes among women from a fertility clinic. Reprod Toxicol. 2015 Jan;51:125-132. doi: 10.1016/j.reprotox.2015.01.003. Epub 2015 Jan 17. PMID 25601638
- [Result] Gaskins AJ, Rich-Edwards JW, Hauser R, Williams PL, Gillman MW, Penzias A, Missmer SA, Chavarro JE. Prepregnancy dietary patterns and risk of pregnancy loss. Am J Clin Nutr. 2014 Oct;100(4):1166-72. doi: 10.3945/ajcn.114.083634. Epub 2014 Aug 13. PMID 25240079
- [Result] Peretz J, Vrooman L, Ricke WA, Hunt PA, Ehrlich S, Hauser R, Padmanabhan V, Taylor HS, Swan SH, VandeVoort CA, Flaws JA. Bisphenol a and reproductive health: update of experimental and human evidence, 2007-2013. Environ Health Perspect. 2014 Aug;122(8):775-86. doi: 10.1289/ehp.1307728. Epub 2014 Jun 4. PMID 24896072
- [Result] Gaskins AJ, Rich-Edwards JW, Hauser R, Williams PL, Gillman MW, Ginsburg ES, Missmer SA, Chavarro JE. Maternal prepregnancy folate intake and risk of spontaneous abortion and stillbirth. Obstet Gynecol. 2014 Jul;124(1):23-31. doi: 10.1097/AOG.0000000000000343. PMID 24901281
- [Result] Meeker JD, Cooper EM, Stapleton HM, Hauser R. Exploratory analysis of urinary metabolites of phosphorus-containing flame retardants in relation to markers of male reproductive health. Endocr Disruptors (Austin). 2013 Oct 1;1(1):e26306. doi: 10.4161/endo.26306. PMID 24795899
- [Result] Meeker JD, Cooper EM, Stapleton HM, Hauser R. Urinary metabolites of organophosphate flame retardants: temporal variability and correlations with house dust concentrations. Environ Health Perspect. 2013 May;121(5):580-5. doi: 10.1289/ehp.1205907. Epub 2013 Mar 5. PMID 23461877
- [Result] Braun JM, Sathyanarayana S, Hauser R. Phthalate exposure and children's health. Curr Opin Pediatr. 2013 Apr;25(2):247-54. doi: 10.1097/MOP.0b013e32835e1eb6. PMID 23429708
- [Result] Johnson PI, Stapleton HM, Mukherjee B, Hauser R, Meeker JD. Associations between brominated flame retardants in house dust and hormone levels in men. Sci Total Environ. 2013 Feb 15;445-446:177-84. doi: 10.1016/j.scitotenv.2012.12.017. Epub 2013 Jan 16. PMID 23333513
- [Result] McAuliffe ME, Williams PL, Korrick SA, Dadd R, Perry MJ. The association between sperm sex chromosome disomy and semen concentration, motility and morphology. Hum Reprod. 2012 Oct;27(10):2918-26. doi: 10.1093/humrep/des302. Epub 2012 Aug 14. PMID 22892419
- [Result] Mendiola J, Meeker JD, Jorgensen N, Andersson AM, Liu F, Calafat AM, Redmon JB, Drobnis EZ, Sparks AE, Wang C, Hauser R, Swan SH. Urinary concentrations of di(2-ethylhexyl) phthalate metabolites and serum reproductive hormones: pooled analysis of fertile and infertile men. J Androl. 2012 May-Jun;33(3):488-98. doi: 10.2164/jandrol.111.013557. Epub 2011 May 19. PMID 21597090
- [Result] McAuliffe ME, Williams PL, Korrick SA, Altshul LM, Perry MJ. Environmental exposure to polychlorinated biphenyls and p,p'-DDE and sperm sex-chromosome disomy. Environ Health Perspect. 2012 Apr;120(4):535-40. doi: 10.1289/ehp.1104017. Epub 2011 Dec 21. PMID 22189045
- [Result] Perry MJ, Chen X, McAuliffe ME, Maity A, Deloid GM. Semi-automated scoring of triple-probe FISH in human sperm: methods and further validation. Cytometry A. 2011 Aug;79(8):661-6. doi: 10.1002/cyto.a.21078. Epub 2011 May 12. PMID 21567938
- [Result] Meeker JD, Yang T, Ye X, Calafat AM, Hauser R. Urinary concentrations of parabens and serum hormone levels, semen quality parameters, and sperm DNA damage. Environ Health Perspect. 2011 Feb;119(2):252-7. doi: 10.1289/ehp.1002238. Epub 2010 Sep 28. PMID 20876036
- [Result] Johnson PI, Stapleton HM, Sjodin A, Meeker JD. Relationships between polybrominated diphenyl ether concentrations in house dust and serum. Environ Sci Technol. 2010 Jul 15;44(14):5627-32. doi: 10.1021/es100697q. PMID 20521814
- [Result] Meeker JD, Stapleton HM. House dust concentrations of organophosphate flame retardants in relation to hormone levels and semen quality parameters. Environ Health Perspect. 2010 Mar;118(3):318-23. doi: 10.1289/ehp.0901332. PMID 20194068
- [Result] Meeker JD, Johnson PI, Camann D, Hauser R. Polybrominated diphenyl ether (PBDE) concentrations in house dust are related to hormone levels in men. Sci Total Environ. 2009 May 1;407(10):3425-9. doi: 10.1016/j.scitotenv.2009.01.030. Epub 2009 Feb 10. PMID 19211133
- [Result] Meeker JD, Calafat AM, Hauser R. Urinary metabolites of di(2-ethylhexyl) phthalate are associated with decreased steroid hormone levels in adult men. J Androl. 2009 May-Jun;30(3):287-97. doi: 10.2164/jandrol.108.006403. Epub 2008 Dec 4. PMID 19059903
- [Result] Meeker JD, Barr DB, Hauser R. Pyrethroid insecticide metabolites are associated with serum hormone levels in adult men. Reprod Toxicol. 2009 Apr;27(2):155-60. doi: 10.1016/j.reprotox.2008.12.012. Epub 2009 Jan 24. PMID 19429394
- [Result] Mahalingaiah S, Meeker JD, Pearson KR, Calafat AM, Ye X, Petrozza J, Hauser R. Temporal variability and predictors of urinary bisphenol A concentrations in men and women. Environ Health Perspect. 2008 Feb;116(2):173-8. doi: 10.1289/ehp.10605. PMID 18288314
- [Result] Meeker JD, Ravi SR, Barr DB, Hauser R. Circulating estradiol in men is inversely related to urinary metabolites of nonpersistent insecticides. Reprod Toxicol. 2008 Feb;25(2):184-91. doi: 10.1016/j.reprotox.2007.12.005. Epub 2007 Dec 28. PMID 18249523
- [Result] Meeker JD, Calafat AM, Hauser R. Di(2-ethylhexyl) phthalate metabolites may alter thyroid hormone levels in men. Environ Health Perspect. 2007 Jul;115(7):1029-34. doi: 10.1289/ehp.9852. PMID 17637918
- [Result] Meeker JD, Altshul L, Hauser R. Serum PCBs, p,p'-DDE and HCB predict thyroid hormone levels in men. Environ Res. 2007 Jun;104(2):296-304. doi: 10.1016/j.envres.2006.11.007. Epub 2006 Dec 26. PMID 17189629
- [Result] Duty SM, Ackerman RM, Calafat AM, Hauser R. Personal care product use predicts urinary concentrations of some phthalate monoesters. Environ Health Perspect. 2005 Nov;113(11):1530-5. doi: 10.1289/ehp.8083. PMID 16263507
- [Result] Chen Z, Godfrey-Bailey L, Schiff I, Hauser R. Impact of seasonal variation, age and smoking status on human semen parameters: The Massachusetts General Hospital experience. J Exp Clin Assist Reprod. 2004 Sep 30;1(1):2. doi: 10.1186/1743-1050-1-2. PMID 15507127
- [Derived] Moyd SA, Hood RB, Zhang Q, Minguez-Alarcon L, Hauser R, Souter I, Gaskins AJ. Maternal and paternal smoking and offspring antral follicle count in women from an infertility clinic. Int J Hyg Environ Health. 2025 Dec 3;272:114719. doi: 10.1016/j.ijheh.2025.114719. Online ahead of print. PMID 41343907
- [Derived] Kadir M, Hood RB, Minguez-Alarcon L, Maldonado-Carceles AB, Ford JB, Souter I, Chavarro JE, Gaskins AJ; EARTH Study Team. Folate intake and ovarian reserve among women attending a fertility center. Fertil Steril. 2022 Jan;117(1):171-180. doi: 10.1016/j.fertnstert.2021.09.037. Epub 2021 Nov 19. PMID 34809974
- [Derived] Nassan FL, Chiu YH, Vanegas JC, Gaskins AJ, Williams PL, Ford JB, Attaman J, Hauser R, Chavarro JE; EARTH Study Team. Intake of protein-rich foods in relation to outcomes of infertility treatment with assisted reproductive technologies. Am J Clin Nutr. 2018 Nov 1;108(5):1104-1112. doi: 10.1093/ajcn/nqy185. PMID 30475972